CLINICAL TRIAL: NCT07399392
Title: Radial Versus Femoral Secondary Access in Patients Undergoing TAVI
Acronym: RADIAL-TAVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Heart Center Freiburg - Bad Krozingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-1058-S1
Record Dates: First submitted 2025-11-27; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: TAVI(Transcatheter Aortic Valve Implantation)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Radial (Active Comparator): Group 1: patients with radial secondary arterial access
  Interventions: Procedure: Radial TAVI
- Group 2 femoral (Active Comparator): Group 2: patients with femoral secondary arterial access
  Interventions: Procedure: femoral TAVI

INTERVENTIONS:
Procedure: Radial TAVI — patients will recieve the TAVI intervention via radial access
  Arms: Group 1 Radial
Procedure: femoral TAVI — patients will recieve the TAVI intervention via femoral access
  Arms: Group 2 femoral

SUMMARY:
Severe symptomatic aortic stenosis (AS) with a high gradient is associated with a poor prognosis if not treated with valve replacement. Transcatheter aortic valve implantation has been shown in large randomized trials to be a safe and effective treatment option for patients at low, intermediate, or high risk. Transfemoral access for heart valve replacement is by far the most commonly used approach, as it is relatively easy to control and has a low complication rate compared to other access routes.

The TAVI procedure requires two arterial access points: one with a large lumen for the TAVI prosthesis via the femoral artery, and a smaller second one for a pigtail catheter that guides the TAVI prosthesis into the optimal position. This secondary access is most often via a second artery.

Vascular complications are the most commonly observed complications in transfemoral TAVI and are associated with poorer procedural outcomes.

Recent data suggest that secondary vascular access via the radial artery may contribute to a reduction in vascular complications after TAVI. In patients undergoing coronary angiography and/or percutaneous coronary intervention, radial access has become the preferred strategy due to its proven reduction in vascular complications compared to femoral access. The use of radial access is associated with a lower incidence of vascular complications compared to femoral access.

Recent non-randomized data suggest that radial access may be a safer alternative to traditional femoral access as a secondary arterial access in transfemoral TAVI. However, non-randomized retrospective comparisons are subject to selection bias and underreporting of complications. Therefore, a prospective randomized trial is needed to evaluate the value of radial access for secondary arterial access in patients undergoing transfemoral TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for transfemoral TAVI
* Heart team agrees on eligibility of TAVI
* Written informed consent
* Age > 18 years

Exclusion Criteria:

* Non accessible radial arteries as judged by the TAVI team
* Non accessible femoral arteries as judged by the TAVI team
* Foreseeable problems to achieve primary transfemoral access (hostile access)
* Hemodynamic instability or cardiogenic shock
* Currently participating in an investigational drug or another device study
* Lack of capability to give informed consent
* Patient refuses TAVI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Vascular and bleeding complications related to the secondary vascular access site | 30 days

SECONDARY OUTCOMES:
Until 30 days after index procedure: | 30 days
  * cardiovascular mortality
  * non-cardiovascular mortality
  * mortality related to vascular and bleeding complications
  * Incidence of new neurological events after randomization
  * Vascular complications at 30 days
  * Bleeding complications at 30 days
  * Incidence of acute kidney injury

CONTACTS AND LOCATIONS:
Locations (1):
- University Heart Center - Deparment for Cardiology and Angiology, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: Yes
Shared IPD from clinical trials used for further scientific research will be stored in a secure processing environment and, depending on the request for secondary use, will be made accessible either as pseudonymised or anonymised datasets.